CLINICAL TRIAL: NCT00543621
Title: An Intervention Program to Control Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Welltech Study
Record Dates: First submitted 2007-10-12; First posted 2007-10-15 (Estimated); Last update posted 2007-10-15 (Estimated); Status verified 2007-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: daily enteral nutritional product and/or behavioral changes

SUMMARY:
Study to evaluate the effectiveness of a structured intervention to improve diabetes control.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* 18-70 adults
* Type 2 Diabetes
* Males and non-pregnant females

Exclusion Criteria:

* Use of exogenous insulin for glucose control
* Use of medications or supplements for weight loss
* Advanced diabetes complications
* Recent history of cardiovascular event

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-05

PRIMARY OUTCOMES:
HbA1c, Fasting blood glucose,blood pressure, weight loss | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jianqin Sun, MD, MPH, Principal Investigator — Clinical Nutrition Center, Huadong Hospital
Locations (1):
- Huandong Hospital, Shanghai, China